CLINICAL TRIAL: NCT02027285
Title: Nutritional Trial With Fortified Milk in 65+ Years Old Subjects
Brief Title: Nutrition, Health and Quality of Life: Development of New Formulations of Traditional Products of the "Made in Italy" Diet Optimized for Consumers With an Age Over 50 Years (MIAO 50)
Acronym: MIAO50
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Claudio Franceschi, Professor, University of Bologna
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 00088MI01
Record Dates: First submitted 2013-12-17; First posted 2014-01-06 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Aging
Keywords: fortified milk, aging, health status

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- fortified milk (Experimental): The subjects assumed daily 250 ml of fortified milk for 12 weeks. Then, after a period of wash-out of 12-14 weeks they start to assume placebo milk for 12 weeks.
  Interventions: Dietary Supplement: fortified milk
- placebo milk (Placebo Comparator): The subjects assumed daily 250 ml of placebo milk. Then, after a period of wash-out of 12-14 weeks they start to assume fortified milk for 12 weeks.
  Interventions: Dietary Supplement: fortified milk

INTERVENTIONS:
Dietary Supplement: fortified milk — "Fortified"Ultra-high temperature (UHT), partly-skimmed milk (1.6% fat), highly digestible (lactose <0.5%) produced by Granarolo s.p.a. supplemented with long chain unsaturated fatty acids DHA (Docosahexaenoic acid) +EPA (Eicosapentaenoic acid), vitamin D, B12, B6, B9, E,C, Zinc and Selenium versus "placebo" Ultra-high temperature (UHT), partly-skimmed milk (1.6% fat), highly digestible (lactose <0.5%) of the same manufacturer.
  The nutrients added are: DHA + EPA 1.4 mg/ml; vitamin D3 0.068 mcg/ml; B6 6.4 mcg/ml; B12 0.01 mcg/ml; B9 (folic acid) 0.80 mcg/ml; vitamin E 0.05 mg/ml; vitamin C 0.19 mg/ml; Zinc 0.04 mg/ml; Selenium 0.22 mcg/ml. The protein content of the milk is 0.04 g/ml.

SUMMARY:
The study ""Nutritional trial with fortified milk in 65+ years old subjects" is a part of a complex research project and multi-sectoral development (MIAO 50) with the participation of University Research Institutes and small and medium Italian enterprises.

The general objective of the call is to promote the collaboration between the best scientific knowledge, both epidemiological and experimental, and the most advanced technologies to develop foods with a nutritional profile adequate to the needs of consumers with an age over 50 years old, which are easy to use and make it possible to eat in a healthy manner, complete and balanced and also meets the quality and flavors of traditional Italian.

DETAILED DESCRIPTION:
Aging is associated with a functional decline of most physiological systems including the immune system. It could be hypothesized that an inadequate nutritional status may amplify the effects of a low-grade chronic inflammation associated with age influencing the functionality of the immune systems, the resistance to infections, the cognitive function and contributing to an increased morbidity and mortality. Indeed experimental evidence indicate that improving the nutritional status attenuates the decline in immune and cognitive functions, in physical performance associated with age by helping to improve the level of Quality of Life.

Therefore, the present study focus on nutrients and micronutrient which have a role in fighting oxidative stress, in the regulation of inflammatory responses and the immune system.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with an age between 63 and 80 years old, males and females, free-living, resident in Bologna and its province.

Exclusion Criteria:

* Allergy or intolerance to cow's milk or a dislike. Dietary treatments and use of specific supplements of molecules associated with the proposed intervention up to two months before the start of the trial. Presence of celiac disease and other malabsorption. Presence of disease with poor prognosis in the short term. Chronic therapy with anticoagulants, corticosteroids, and anti-cancer. Exclusion of subjects with onset of chronic-degenerative diseases in the last year, presence of type I diabetes and chronic viral hepatitis.

Ages: 63 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Global health status | Change from baseline global health status at 12 weeks of milk intake
  The health status is evaluated by a tests regarding the cognitive function, the functional status, the perceived health status.

SECONDARY OUTCOMES:
Circulating levels of lipoproteins (Total, HDL and LDL-cholesterol, triglycerides) | change from baseline total, HDL, and LDL-cholesterol and triglycerides at 12 weeks of milk intake
  total cholesterol is measured as milligram/100milliliters (mg/100ml); HDL-cholesterol as milligram/100milliliters (mg/100ml); LDL-cholesterol as milligram/100milliliters (mg/100ml); triglycerides as milligram/100milliliters (mg/100ml).
Levels of blood glucose, creatinine, liver transaminases, homocysteine, folic acid | Change from Baseline levels of glucose, creatinine, liver transaminases, homocysteine and folic acid at 12 weeks of milk intake
  Glucose was measured as milligram/deciliter (mg/dl); creatinine as milligram/deciliter (mg/dl), liver transaminases as International units/liter (U/L); homocysteine as micromoles/L and folic acid as nanogram/milliliter (ng/ml)
Circulating levels of vitamin D, vitamin E, vitamin B6 and vitamin B12 | Change from Baseline levels of vitamin D, vitamin E, vitamin B6 and vitamin B12 at 12 weeks of milk intake
  Vitamin D was measured as nanogram/milliliters (ng/ml); vitamin E as micrograms/milliliters (mcg/ml); vitamin B6 as micrograms/liter (mcg/L) and vitamin B12 as picograms/milliliters (pg/ml)
Fatty acid composition of red blood cell membranes as an index of cellular homeostasis | Change from Baseline fatty acid composition of red blood cell membranes at 12 weeks of milk intake
Circulating levels of trace elements such as zinc and selenium | Changes from Baseline levels of zinc and selenium at 12 weeks of milk intake
  Zinc and selenium were measured as microgram/liter (mcg/L)
Oxidation state of cellular proteins | Change from Baseline oxidation state of cellular proteins at 12 weeks of milk intake
Circulating levels of proteins related to inflammatory status such as C reactive protein (CRP); fibrinogen and pro and anti-inflammatory cytokines. | Changes from baseline CRP, fibrinogen, high sensitivity interleukin 6 (hs-IL6) and high sensitivity interleukin 10 (hs-IL10)
  C reactive protein was measured as milligram/liter (mg/l); fibrinogen as milligram/deciliter (mg/dl); hs-IL6 and hs-IL10 as picograms/milliliter (pg/ml)
Blood count and assessment of major lymphocyte sub-populations | Change from Baseline lymphocyte subsets at 12 weeks of milk intake

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Franceschi, MD, Study Chair — University of Bologna
Locations (1):
- University of Bologna-Department of Speciality, Diagnostic and Experimental Medicine, Bologna, Bologna, Italy